CLINICAL TRIAL: NCT03647228
Title: A Double-Blind, Placebo-Controlled, Dose-Escalation, Phase 1/2a Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single and Multiple Doses of ION-827359, an Antisense Oligonucleotide Inhibitor of ENaC, Administered to Healthy Volunteers and Patients With Cystic Fibrosis
Brief Title: A Phase 1/2a Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single and Multiple Doses of IONIS-ENaCRx in Healthy Volunteers and Patients With Cystic Fibrosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ionis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ION-827359-CS1; 2018-002621-27 (EudraCT Number)
Record Dates: First submitted 2018-08-23; First posted 2018-08-27 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Healthy Subjects; Cystic Fibrosis
Keywords: ION-827359; ENaC
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- IONIS-ENaCRx (Experimental): Ascending single and multiple doses of IONIS-ENaCRx inhaled or nebulized.
  Interventions: Drug: IONIS-ENaCRx
- Placebo (Placebo Comparator): Placebo comparator calculated volume to match active comparator inhaled or nebulized.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: IONIS-ENaCRx — Ascending single and multiple doses of IONIS-ENaCRx inhaled or nebulized.
  Arms: IONIS-ENaCRx
Drug: Placebo — Placebo comparator calculated volume to match active comparator inhaled or nebulized.
  Arms: Placebo

SUMMARY:
This Phase 1/2a study is a double-blinded (subject and Investigator), randomized, placebo-controlled, dose-escalation study to evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of single and multiple nebulized doses of IONIS-ENaCRx.

DETAILED DESCRIPTION:
This study will be conducted in 3 parts: a single ascending dose (SAD) leading to a multiple ascending dose (MAD) in healthy volunteers, followed by a MAD in patients with cystic fibrosis. The study will enroll up to 88 participants.

The study will consist of 4 single-dose randomized cohorts. Participants enrolled will receive a single inhaled dose of the Study Drug (IONIS-ENaCRx or placebo) on Day 1.

ELIGIBILITY:
Inclusion Criteria (Healthy Volunteers)

1. Females must be non-pregnant and non-lactating, and either surgically sterile or post-menopausal.
2. Males must be surgically sterile or, abstinent or, if engaged in sexual relations with a woman of child-bearing potential, the subject or the subject's non-pregnant female partner must be using a highly effective contraceptive method
3. Willing to refrain from strenuous exercise/activity for at least 72 hours prior to study visits
4. Body mass index (BMI) < 35 kg/m2 with a minimum weight of 45 kg
5. Normal diffusing capacity in the lung (≥ 80% predicted) at Screening

Exclusion Criteria (Healthy Volunteers)

1. Clinically-significant (CS) abnormalities in medical history, screening laboratory results, physical or physical examination that would render a subject unsuitable for inclusion, including but not limited to:

   1. Urine protein/creatinine (P/C) ratio ≥ 0.2 mg/mg
   2. Positive test (including trace) for blood on urinalysis
   3. Alanine aminotransferase (ALT), aspartate aminotransferase (AST), bilirubin, alkaline phosphatase (ALP), serum creatinine, blood urea nitrogen (BUN), fasting blood glucose, potassium > upper limit of normal (ULN)
   4. Platelet count < LLN
2. Active infection requiring systemic antiviral or antimicrobial therapy that will not be completed prior to Study Day 1
3. Respiratory infection within 4 weeks of Study Day 1
4. Presence or past history of CS chronic respiratory disease, including any current history (or within 2 years) of asthma. History of allergic rhinitis is acceptable
5. Forced expiratory volume in 1 second (FEV1) < 80% of predicted at Screening or an FEV1/FVC ratio of < 0.7
6. Smoking of a tobacco or nicotine-containing product within the previous 6 months (use of a nicotine patch is permitted) or a smoking history of ≥ 10 pack years
7. Any CS finding on chest radiograph
8. Uncontrolled hypertension (blood pressure [BP] > 160/100 mm Hg) at Screening
9. Treatment with another investigational drug, biological agent, or device within one month of screening, or 5 half-lives of investigational agent, whichever is longer
10. Any history of previous treatment with an oligonucleotide
11. Regular use of alcohol within 6 months prior to screening or hard drugs within 1 year prior to screening, or positive urine drug screen at Screening
12. Blood donation of 50 to 499 mL within 30 days of screening or of > 499 mL within 60 days of screening

Inclusion Criteria (Cystic Fibrosis Participants)

1. Females must be non-pregnant and non-lactating, and either surgically sterile or post-menopausal.
2. Males must be surgically sterile or, abstinent or, if engaged in sexual relations with a woman of child-bearing potential, the subject or the subject's non-pregnant female partner must be using a highly effective contraceptive method
3. Confirmed diagnosis of CF by seat chloride and/or genetics by referring clinician
4. FEV1 >/= 50% of predicted
5. Stable CF disease as judged by the Investigator
6. Weight > 40 kg

Exclusion Criteria (Cystic Fibrosis Participants)

1. Clinically-significant (CS) abnormalities in medical history, screening laboratory results, physical or physical examination that would render a subject unsuitable for inclusion, including but not limited to:

   1. Abnormal liver function defined as > 2 times upper limit of normal (ULN) for bilirubin, or 3 time ULN for ALT, AST, or alkaline phosphatase
   2. Platelet count < LLN
2. Active infection requiring systemic antiviral or antimicrobial therapy that will not be completed prior to Study Day 1
3. Respiratory infection within 4 weeks of Study Day 1
4. Colonization with Burkholderia cepacia or M. abscessus

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 98 (Actual)
Dates: Start 2018-12-13 (Actual); Primary Completion 2020-10-13 (Actual); Study Completion 2020-10-13 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability as Measured by the Number of Participants with at least one Treatment-Emergent Adverse Event | Up to 113 Days

SECONDARY OUTCOMES:
Cmax: maximum observed drug concentration in plasma of IONIS-ENaCRx | Up to 113 Days
Tmax: time taken to reach maximal concentration in plasma of IONIS-ENaCRx | Up to 113 Days
AUCt: area under the plasma concentration-time curve from time zero to time t for IONIS-ENaCRx | Up to 113 Days
CL/F: apparent total clearance of IONIS-ENaCRx | Up to 113 Days
t1/2λz: termination half-life of IONIS-ENaCRx | Up to 113 Days
The amount of administered dose of IONIS-ENaCRx excreted in urine over a 24-hour period | Up to 113 Days

CONTACTS AND LOCATIONS:
Locations (8):
- Germany (3):
  - Universitätsmedizin Essen, Essen
  - Universitätsklinikum Frankfurt, Frankfurt
  - Lungenheilkunde München-Pasing, München
- United Kingdom (5):
  - Medicines Evaluation Unit, Wythenshawe, Manchester
  - Celerion, Belfast, Northern Ireland
  - Western General Hospital, Edinburgh
  - Adults Cystic Fibrosis King's College Hospital - Hambleden Wing (East), London
  - Royal Brompton Hospital, London

IPD SHARING:
Plan to Share IPD: No